CLINICAL TRIAL: NCT02316002
Title: Phase II Study of Pembrolizumab After Curative Intent Treatment for Oligometastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 25514
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Oligometastatic Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg every 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab

SUMMARY:
The main purpose of this study is to see how well the experimental drug pembrolizumab (MK-3475) works in people with oligometastatic NSCLC who have already had treatment for their disease. All patients will receive 200 mg of pembrolizumab intravenously on Day 1 of each 21-day cycle. Patients will receive the study drug for up to 8 cycles, and then if their disease is doing well and the study doctor thinks they will benefit patients may receive pembrolizumab for up to 8 more cycles.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent for the trial.
* 18 years of age on day of signing informed consent.
* Completion of definitive therapy 4-12 weeks prior to enrollment. There are no specific limitations on which treatment modalities can be used in the definitive setting (e.g. the use of adjuvant chemotherapy is acceptable), but all other treatments must be complete at least 4 weeks prior to enrollment.
* Provision of tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion.

  1. Tumor tissue may be from a diagnostic biopsy or a portion of a surgical specimen, if surgery is a component of definitive intent therapy.
  2. Formalin fixed paraffin embedded (FFPE) tissue samples are acceptable; a fine needle aspirate, frozen sample, plastic embedded sample, cell block, clot, bone, bone marrow or cytologic specimen will not be acceptable for IHC analysis.
  3. It is recommended that FFPE blocks be sectioned fresh (within 7 days of sectioning and sending for PD-L1 analysis) onto positively charged slides; slides should be stored and shipped (and stored upon receipt at Qualtek) at 2-8C in the dark.
  4. Recommended fixation time for samples is 24 hours to 48 hours in 10% neutral buffered formalin.
* Performance status of 0 or 1 on the ECOG Performance Scale.
* Adequate organ function, all screening labs should be performed within 10 days of treatment initiation.

Absolute neutrophil count

* 1,250 /mcL Product: Pembrolizumab Protocol/Amendment No.: 09/19/2014 10 (ANC) Platelets
* 100,000 / mcL Hemoglobin
* 9 g/dL or ≥5.6 mmol/L Renal Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl)

  ≤1.5 X upper limit of normal (ULN) OR
* 50 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin

  * 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT)
  * 2.5 X ULN OR
  * 5 X ULN for subjects with liver metastases aCreatinine clearance should be calculated per institutional standard.

    * Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
    * Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the duration of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
    * Male subjects who are partnered with women of childbearing potential should be willing to use 2 methods of birth control, be surgically sterile or abstain from heterosexual activity for the duration of the study through 120 days after the last dose of study medication.

Exclusion Criteria:

* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Diagnosis of immunodeficiency or exposure to systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (Nasal or oral inhalers are permissible).
* Prior monoclonal antibody within 4 weeks prior to study Day 1 or individuals who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Day 1 drug administration on study or inability to recover (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy or alopecia are exceptions to this criterion and may qualify for the study.
* Note: If subject had major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, non-invasive bladder tumors, or in situ cervical cancer
* Known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome are not excluded from the study.
* Evidence of pre-existing interstitial lung disease or active, non-infectious pneumonitis.
* Active infection requiring systemic therapy with IV antibiotics
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg positive or HBV DNA detectable) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Receipt of live vaccine within 30 days prior to the first dose of trial treatment.
* Progressive disease or sites of new metastasis after definitive therapy for oligometastatic disease.
* Completion of definitive therapy for oligometastatic disease greater than 12 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bauml JM, Mick R, Ciunci C, Aggarwal C, Davis C, Evans T, Deshpande C, Miller L, Patel P, Alley E, Knepley C, Mutale F, Cohen RB, Langer CJ. Pembrolizumab After Completion of Locally Ablative Therapy for Oligometastatic Non-Small Cell Lung Cancer: A Phase 2 Trial. JAMA Oncol. 2019 Sep 1;5(9):1283-1290. doi: 10.1001/jamaoncol.2019.1449. PMID 31294762

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Pembrolizumab 200 mg every 3 weeks
  Pembrolizumab
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 51
Completed | 45
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 64 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time to progression or death from initiation of LAT
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 45
Months | 19.1 [9.4 to 28.7]

ADVERSE EVENTS:
Time Frame: 2 years
Description: As per CTCAE
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 11/45
Serious Adverse Events (participants affected / at risk) | 15/45
Other Adverse Events (participants affected / at risk) | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=45)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02316002/Prot_SAP_000.pdf